CLINICAL TRIAL: NCT06400069
Title: Evaluation of Serum NLRP6 in Chronic Periodontitis Patients
Brief Title: Role of NLRP6 in Chronic Periodontitis
Status: Completed | Type: Observational
Sponsor: Babol University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Morteza Rabbani, Morteza Rabbani, DS, Babol University of Medical Sciences
Other Study IDs: IR.MUBABOL.REC.1403.037
Record Dates: First submitted 2024-04-30; First posted 2024-05-06 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-04

CONDITIONS: Chronic Periodontitis
Keywords: NLRP6 Protein, human; Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Evaluation of serum NLRP6 levels — intervention: Evaluation of serum NLRP6 levels control: Evaluation of serum NLRP6 levels

SUMMARY:
The quantification of NLRP6 in blood samples will be analyzed from individuals with chronic periodontitis but without systemic disease. Demographic and periodontal parameters will be assessed and correlated with the NLRP6 quantification using RT-PCR.

DETAILED DESCRIPTION:
This study aims to collect demographic variables, including age, education level, BMI, personal habits, medication use, and history of systemic disease, from non-smoking individuals with chronic periodontitis. Initially, we will determine the expression level of the NLRP6 gene in blood samples taken from chronic periodontitis subjects who are matched for age and sex. Subsequently, we will investigate the relationship between gene expression levels, taking into account the confounding effect of body mass index, and explore how these levels correlate with the severity of the disease.

In this study, two groups: chronic periodontitis (CP) and healthy controls (HC) will be examined. The CP group will consist of patients diagnosed with Stage I to IV periodontitis based on the consensus report from the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. Additionally, we will include systemically healthy individuals. Serum samples will be collected from all patients, and the Plaque Index (PI) and Gingival Index (GI) will be recorded at four sites per tooth. Furthermore, we will assess full-mouth probing depth (PD) and clinical attachment level (CAL) at six sites per tooth. The percentage of bleeding areas will be documented as the proportion of sites with bleeding on probing (BOP) within 20 seconds after probing.

For blood sampling, a total of 3 mL of blood will be collected from the antecubital vein of each individual by an expert nurse from the Department of Periodontology.

Statistical analysis will be conducted using statistical software for data science (Stata version 17). A significance value (p-value) of less than 0.05 will be considered statistically significant. The sample size for the study was determined using the power paired means module in Stata 17. We planned to include at least 25 individuals in each group, aiming for a significance level of 5%, statistical power of 80%, and a correlation coefficient of 0.2.

ELIGIBILITY:
Inclusion Criteria:

* Age: At least 25 years old
* Clinical diagnosis of chronic periodontitis
* At least 15 teeth in the mouth

Exclusion Criteria:

* premalignant lesions and cancer of the oral cavity
* periodontal treatment in the last 6 months
* systemic disorders affecting the periodontal condition (autoimmunity and endocrine disorders)
* diabetes mellitus and rheumatoid arthritis
* pregnancy or breastfeeding
* taking drugs with the possibility of affecting the periodontal condition (calcium channel blockers, anticonvulsants, etc.)
* Smoking
* aggressive PD

Ages: 25 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to the periodontology department of the University School of Dentistry Medical sciences of Babol
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2024-12-13 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-11-22 (Actual)

PRIMARY OUTCOMES:
Quantification of NLRP6 gen, Quantification of NLRP6 gen using RT-PCR | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Dental School, Periodontology Department, Babol, Iran

IPD SHARING:
Plan to Share IPD: Undecided